CLINICAL TRIAL: NCT00466258
Title: LINFOTARGAM: First-line Treatment With Dose-dense Chemotherapy Plus Rituximab (R-CHOP/14) and Highly Active Antiretroviral Therapy (HAART) in Patients With Diffuse Large B Cell Lymphoma (DLBCL) and Infection With the Human Immunodeficiency Virus (HIV)
Brief Title: LINFOTARGAM: Treatment With Chemotherapy Plus Rituximab and Highly Active Antiretroviral Therapy in Patients With Diffuse Large B Cell Lymphoma and Infection With the Human Immunodeficiency Virus (HIV)
Acronym: LINFOTARGAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-003750-23; LINFOTARGAM
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infections; Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B cell lymphoma; HIV; R-CHOP; Highly active antiretroviral therapy; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Antiretroviral Therapy, Highly Active; Nurse Clinicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: R-CHOP — * Cyclophosphamide 750 mg/m2 i.v. day 1
  * Adriamycin 50 mg/m2 i.v. day 1
  * Vincristine 1,4 mg/m2 i.v. day 1
  * Prednisone 100 mg i.v or oral. days 1-5.
Drug: Highly active antiretroviral therapy — Combined antiretroviral treatment (TARGA) wich include at lest 3 drugs. The combination should be accepted as an initial or rescue treatment.
Drug: Central nervous system (CNS) prophylaxis — methotrexate (12 mg) cytarabine (30 mg) hydrocortisone (20 mg)
Drug: Prophylaxis of opportunistic infections and support treatment — Pegfilgrastim

SUMMARY:
Main objective:

* To evaluate the applicability of the treatment:

  1. To evaluate the treatment toxicity according to the Common Terminology Criteria (CTC) version 3.0 of the National Cancer Institute (NCI).
  2. To evaluate opportunistic and non-opportunistic infections after 6 cycles of treatment with rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) administered every 14 days and highly active antiretroviral therapy (HAART) in patients with diffuse large B cell lymphoma (DLBCL) and HIV infection.
  3. To evaluate the adherence to the treatment with 6 cycles of R-CHOP considering the delays in the administration of the cycles and the reductions in the doses of chemotherapy (planned dose administered in predicted term).

Secondary objectives:

* To evaluate the efficacy of the treatment in patients with DLBCL and HIV infection after 6 cycles of treatment with R-CHOP administered every 14 days (R-CHOP/14):

  1. To determine the global response and complete remission tax.
  2. To evaluate the duration of the response.
  3. To evaluate the probability of event-free survival in 5 years.
  4. To evaluate the probability of global survival in 5 years.
* To identify predictive factors of response after 6 cycles of treatment with R-CHOP administered every 14 days in patients with DLBCL and HIV infection.
* To evaluate the impact of the therapeutic combination of R-CHOP and HAART in the parameters of the HIV infection (HIV viral load and CD4+ lymphocyte count).

DETAILED DESCRIPTION:
This is a clinical trial with a pharmaceutical drug used in the same conditions of authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV infection diagnosed with DLBCL in any stage (I-IV according to the Ann Arbor classification) not previously treated for the lymphoma.
* Patients with CD20-positive diffuse large B-cell lymphoma
* Aged from 18 to 70 years old
* Any score of International Prognostic Index. (It is also applicable in patients with non-Hodgkin lymphoma [NHL] infected with HIV.)
* ECOG performance status 0 to 3
* Written informed consent
* Absolute neutrophil count > 1.5 x 10^9/L.
* Absence of synchronic or non-synchronic neoplasia with the exception of non-melanoma skin tumors or in situ cervical carcinoma.
* CD4+ lymphocyte count > 100/µL

Exclusion Criteria:

* Patients with diffuse large B cell lymphoma previously treated.
* Patients with primary central nervous system lymphoma.
* Patients with Burkitt or Burkitt-like NHL.
* CD4+ lymphocyte count < 100/µL
* Opportunistic infections or other AIDS-related neoplasias in activity.
* Active drug-addiction.
* Pregnant or lactating women or adults of fertile age who do not use an effective contraceptive method.
* Patients with serious altered renal function (creatinine > 2.5 x upper limit of normal [ULN]) or hepatic [bilirubin, ALT or AST > 2.5 x ULN], except if the investigators suspect that they are caused by the disease.
* Cardiac insufficiency with ejection fraction < 40%
* Patients with serious psychiatric diseases that can interfere with their capacity to understand the study (including alcoholism or active drug-addiction).
* ECOG > 3
* Patients with a known hypersensitivity to murine proteins or any other component of the study drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
treatment toxicity according to the CTC criteria (version 3.0) of the National Cancer Institute (NCI) | 6 months
opportunistic and non-opportunistic infections rate after 6 cycles of treatment with R-CHOP administered every 14 days and HAART in patients with DLBCL and HIV infection | 6 months
adherence to the treatment with 6 cycles of R-CHOP considering the delays in the administration of the cycles and the reductions in the doses of chemotherapy (planned dose administered in predicted term) | 6 months

SECONDARY OUTCOMES:
efficacy of the treatment in patients with DLBCL and HIV infection after 6 cycles of treatment with R-CHOP administered every 14 days | 1 year
global response and complete remission rate | 1 year
duration of the response | 5 years
event-free survival probability in 5 years | 5 years
global survival probability in 5 years | 5 years
predictive factors of the response after 6 cycles of treatment with R-CHOP administered every 14 days in patients with DLBCL and HIV infection | 2 years
impact of the therapeutic combination of R-CHOP and HAART in the parameters of the HIV infection (HIV viral load and CD4+ lymphocyte count) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep M, Dr, Principal Investigator — Germans Trias i Pujol Hospital; Oriol Albert, Dr, Principal Investigator — Germans Trias i Pujol Hospital
Locations (15):
- Spain (15):
  - H. Son Llatzer, Palma de Mallorca, Balearic Islands
  - Germans Trias i Pujol, Badalona, Barcelona
  - H. Clínic i Provincial, Barcelona, Barcelona, Barcelona
  - H. Vall d'Hebron, Barcelona, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona, Barcelona, Barcelona
  - ICO - Duran i Reynals, Hospitalet de Llobregat, Barcelona, Barcelona
  - Consorci Sanitari de Mataró, Mataró, Barcelona
  - H. Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - ICO - Josep Trueta, Girona, Girona
  - H. Gregorio Marañón, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - H. Joan XXIII, Tarragona, Tarragona
  - Hospital Universitario Dr. Peset, Valencia, Valencia

REFERENCES:
- [Background] Engels EA, Goedert JJ. Human immunodeficiency virus/acquired immunodeficiency syndrome and cancer: past, present, and future. J Natl Cancer Inst. 2005 Mar 16;97(6):407-9. doi: 10.1093/jnci/dji085. No abstract available. PMID 15769998
- [Background] Noy A. Update in HIV-associated lymphoma. Curr Opin Oncol. 2004 Sep;16(5):450-4. doi: 10.1097/00001622-200409000-00007. PMID 15314514
- [Background] Bonnet F, Lewden C, May T, Heripret L, Jougla E, Bevilacqua S, Costagliola D, Salmon D, Chene G, Morlat P. Malignancy-related causes of death in human immunodeficiency virus-infected patients in the era of highly active antiretroviral therapy. Cancer. 2004 Jul 15;101(2):317-24. doi: 10.1002/cncr.20354. PMID 15241829
- [Background] Carrieri MP, Pradier C, Piselli P, Piche M, Rosenthal E, Heudier P, Durant J, Serraino D. Reduced incidence of Kaposi's sarcoma and of systemic non-hodgkin's lymphoma in HIV-infected individuals treated with highly active antiretroviral therapy. Int J Cancer. 2003 Jan 1;103(1):142-4. doi: 10.1002/ijc.10790. No abstract available. PMID 12455069
- [Background] Ribera JM, Navarro JT. [Lymphomas in patients with HIV infection. A change for the better]. Enferm Infecc Microbiol Clin. 2004 Jun-Jul;22(6):313-4. doi: 10.1157/13063040. No abstract available. Spanish. PMID 15228895
- [Background] Hoffmann C, Chow KU, Wolf E, Faetkenheuer G, Stellbrink HJ, van Lunzen J, Jaeger H, Stoehr A, Plettenberg A, Wasmuth JC, Rockstroh J, Mosthaf F, Horst HA, Brodt HR. Strong impact of highly active antiretroviral therapy on survival in patients with human immunodeficiency virus-associated Hodgkin's disease. Br J Haematol. 2004 May;125(4):455-62. doi: 10.1111/j.1365-2141.2004.04934.x. PMID 15142115
- [Background] Navarro JT, Lloveras N, Ribera JM, Oriol A, Mate JL, Feliu E. The prognosis of HIV-infected patients with diffuse large B-cell lymphoma treated with chemotherapy and highly active antiretroviral therapy is similar to that of HIV-negative patients receiving chemotherapy. Haematologica. 2005 May;90(5):704-6. PMID 15921395
- [Background] Spina M, Carbone A, Vaccher E, Gloghini A, Talamini R, Cinelli R, Martellotta F, Tirelli U. Outcome in patients with non-hodgkin lymphoma and with or without human immunodeficiency virus infection. Clin Infect Dis. 2004 Jan 1;38(1):142-4. doi: 10.1086/380129. Epub 2003 Dec 5. PMID 14679461
- [Background] J Berenguer, R Rubio, JM Ribera, A Antela, J Santos, P Miralles, et al. 10Th Congress of Retroviruses and Opportunistic infections. 2003. Characteristics and outcome of AIDS-related non-Hodgkin's lymphoma before and alter the introduction of HAART (GESIDA 23/01). Abstract 802
- [Background] Simonelli C, Spina M, Cinelli R, Talamini R, Tedeschi R, Gloghini A, Vaccher E, Carbone A, Tirelli U. Clinical features and outcome of primary effusion lymphoma in HIV-infected patients: a single-institution study. J Clin Oncol. 2003 Nov 1;21(21):3948-54. doi: 10.1200/JCO.2003.06.013. PMID 14581418
- [Background] Pantanowitz Lbeckwith B, Dezube BJ. HIV-associated plasma cell neoplasia. HIV AIDS Rev 2004; 3: 47-50.
- [Background] Mate JL, Navarro JT, Ariza A, Ribera JM, Castella E, Junca J, Tural C, Nomdedeu JF, Bellosillo B, Serrano S, Granada I, Milla F, Feliu E. Oral solid form of primary effusion lymphoma mimicking plasmablastic lymphoma. Hum Pathol. 2004 May;35(5):632-5. doi: 10.1016/j.humpath.2003.11.005. PMID 15138941
- [Background] Navarro JT, Ribera JM, Junca J, Milla F. Anorectal lymphoma without effusion associated with human herpesvirus-8 and type 1 Epstein-Barr virus in an HIV-infected patient. Hum Pathol. 2003 Jun;34(6):630. doi: 10.1016/s0046-8177(03)00093-5. No abstract available. PMID 12827623
- [Background] Skiest DJ, Crosby C. Survival is prolonged by highly active antiretroviral therapy in AIDS patients with primary central nervous system lymphoma. AIDS. 2003 Aug 15;17(12):1787-93. doi: 10.1097/00002030-200308150-00007. PMID 12891064
- [Background] JM Ribera, A Oriol, M Morgades, E Gonzalez-Barca, A López-Guillermo, A López, et al. Treatment with rituximab, CHOP and highly active antiretroviral therapy (HAART) in AIDS-related diffuse large B-cell lymphomas (DLBCL). Study of 60 patients. American Society of Hematology. 47th Annual Meeting. Atlanta, December 10-13, 2005. Abstract 774. Blood 2005, 106 (11): 228a.
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Pfreundschuh M, Trumper L, Kloess M, Schmits R, Feller AC, Rudolph C, Reiser M, Hossfeld DK, Metzner B, Hasenclever D, Schmitz N, Glass B, Rube C, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group. Two-weekly or 3-weekly CHOP chemotherapy with or without etoposide for the treatment of young patients with good-prognosis (normal LDH) aggressive lymphomas: results of the NHL-B1 trial of the DSHNHL. Blood. 2004 Aug 1;104(3):626-33. doi: 10.1182/blood-2003-06-2094. Epub 2004 Feb 24. PMID 14982884
- [Background] Pfreundschuh M, Trumper L, Kloess M, Schmits R, Feller AC, Rube C, Rudolph C, Reiser M, Hossfeld DK, Eimermacher H, Hasenclever D, Schmitz N, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group. Two-weekly or 3-weekly CHOP chemotherapy with or without etoposide for the treatment of elderly patients with aggressive lymphomas: results of the NHL-B2 trial of the DSHNHL. Blood. 2004 Aug 1;104(3):634-41. doi: 10.1182/blood-2003-06-2095. Epub 2004 Mar 11. PMID 15016643
- [Background] Tanosaki R, Okamoto S, Akatsuka N, Ishida A, Michikawa N, Masuda Y, Uchida H, Murata M, Kizaki M, Ikeda Y. Dose escalation of biweekly cyclophosphamide, doxorubicin, vincristine, and prednisolone using recombinant human granulocyte colony stimulating factor in non-Hodgkin's lymphoma. Cancer. 1994 Oct 1;74(7):1939-44. doi: 10.1002/1097-0142(19941001)74:73.0.co;2-c. PMID 7521788
- [Background] Grigg A, Solal-Celigny P, Hoskin P, Taylor K, McMillan A, Forstpointner R, Bacon P, Renwick J, Hiddemann W; International Study Group. Open-label, randomized study of pegfilgrastim vs. daily filgrastim as an adjunct to chemotherapy in elderly patients with non-Hodgkin's lymphoma. Leuk Lymphoma. 2003 Sep;44(9):1503-8. doi: 10.1080/1042819031000103953. PMID 14565651
- [Background] Lopez A, Fernandez de Sevilla, A, Castaigne S, Greil R, Sierra J, Sanchez J, et al. Pegfigrastim supports delivery of CHOP-R chemotherapy administered every 14 days: a randomised phase II study. Blood 2004; 104: 904a-905a (abstract 3311).
- [Background] Spina M, Jaeger U, Sparano JA, Talamini R, Simonelli C, Michieli M, Rossi G, Nigra E, Berretta M, Cattaneo C, Rieger AC, Vaccher E, Tirelli U. Rituximab plus infusional cyclophosphamide, doxorubicin, and etoposide in HIV-associated non-Hodgkin lymphoma: pooled results from 3 phase 2 trials. Blood. 2005 Mar 1;105(5):1891-7. doi: 10.1182/blood-2004-08-3300. Epub 2004 Nov 18. PMID 15550484
- [Background] Boue F, Gabarre J, Gisselbrecht Ch, Reynes J, Plantier I, Morlat P, et al. CHOP chemotherapy plus rituximab in HIV patients with high-grade lymphoma. Results of an ANRS trial. 44th Annual Meeting of the American Society of Hematology 2002. Blood 2002; 100 (suppl): 470a.
- [Background] Kaplan LD, Lee JY, Ambinder RF, Sparano JA, Cesarman E, Chadburn A, Levine AM, Scadden DT. Rituximab does not improve clinical outcome in a randomized phase 3 trial of CHOP with or without rituximab in patients with HIV-associated non-Hodgkin lymphoma: AIDS-Malignancies Consortium Trial 010. Blood. 2005 Sep 1;106(5):1538-43. doi: 10.1182/blood-2005-04-1437. Epub 2005 May 24. PMID 15914552
- [Background] Oriol A, Ribera JM, Esteve J, Sanz MA, Brunet S, Garcia-Boyero R, Fernandez-Abellan P, Marti JM, Abella E, Sanchez-Delgado M, Penarrubia MJ, Besalduch J, Moreno MJ, Borrego D, Feliu E, Ortega JJ; PETHEMA Group, Spanish Society of Hematology. Lack of influence of human immunodeficiency virus infection status in the response to therapy and survival of adult patients with mature B-cell lymphoma or leukemia. Results of the PETHEMA-LAL3/97 study. Haematologica. 2003 Apr;88(4):445-53. PMID 12681972
- [Background] Oriol A, Ribera JM, Brunet S, del Potro E, Abella E, Esteve J. Highly active antiretroviral therapy and outcome of AIDS-related Burkitt's lymphoma or leukemia. Results of the PETHEMA-LAL3/97 study. Haematologica. 2005 Jul;90(7):990-2. PMID 15996943
- [Background] Thomas DA, Cortes J, Giles FJ, Faderl S, O'Brien S, Garcia-Manero G, et al. Rituximab and hyper-CVAD for adult Burkitt's or Burkitt-like leukemia or lymphoma. 44th Annual Meeting of the American Society of Hematology 2002. Blood 2002; 100 Suppl 763a.
- [Background] Bokemeyer C, Aapro MS, Courdi A, Foubert J, Link H, Osterborg A, Repetto L, Soubeyran P. EORTC guidelines for the use of erythropoietic proteins in anaemic patients with cancer. Eur J Cancer. 2004 Oct;40(15):2201-16. doi: 10.1016/j.ejca.2004.07.015. PMID 15454245
- [Background] Miralles P, Rubio C, Berenguer J, Ribera JM, Calvo F, Diaz Mediavilla J, Diez-Martin JL, Lopez Aldeguer J, Valencia E, Rubio R. [GESIDA/PETHEMA guidelines for the diagnosis and treatment of lymphomas in HIV-infected patients]. Med Clin (Barc). 2002 Feb 23;118(6):225-36. doi: 10.1016/s0025-7753(02)72342-7. No abstract available. Spanish. PMID 11864547
- [Background] Juweid ME, Wiseman GA, Vose JM, Ritchie JM, Menda Y, Wooldridge JE, Mottaghy FM, Rohren EM, Blumstein NM, Stolpen A, Link BK, Reske SN, Graham MM, Cheson BD. Response assessment of aggressive non-Hodgkin's lymphoma by integrated International Workshop Criteria and fluorine-18-fluorodeoxyglucose positron emission tomography. J Clin Oncol. 2005 Jul 20;23(21):4652-61. doi: 10.1200/JCO.2005.01.891. Epub 2005 Apr 18. PMID 15837965
- See also: Spanish Association of Haematology — http://www.aehh.org